CLINICAL TRIAL: NCT03619408
Title: Management of Esophagitis Following Repair of Esophageal Atresia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Michael A. Manfredi, MD, Assistant Professor of Pediatrics, Harvard Medical School, Boston Children's Hospital
Other Study IDs: P00029371
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Esophageal Atresia; Esophagitis
Keywords: Esophageal Atresia; Esophagitis; GER; Gastroesopheal reflux; PPI
MeSH Terms: conditions — Esophageal Atresia; Esophagitis | interventions — Antacids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — esophageal biopsies obtained with cold forceps during routine surveillance endoscopies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No/Mild Esophagitis: All repaired esophageal atresia patients at Boston Children's Hospital with primary esophageal anastomosis undergoing routine year-1 surveillance endoscopy / pH-impedance studies found to have no or mild histologic esophagitis, no erosive esophagitis, and reflux index <3% on pH-metry. Antacid therapy will be discontinued.
- Moderate/Severe Esophagitis: All repaired esophageal atresia patients at Boston Children's Hospital with primary esophageal anastomosis undergoing routine year-1 surveillance endoscopy / pH-impedance studies found to have moderate or severe histologic esophagitis, and/or erosive esophagitis, and/or reflux index > 3% on pH-metry.
  Antacid therapy with PPI (omeprazole 1mg/kg/dose BID) will be initiated. For patients already taking PPI at therapeutic dosing, an H2 blocker (ranitidine 3mg/kg/dose BID) will be added.
  Interventions: Drug: Antacids

INTERVENTIONS:
Drug: Antacids — Omeprazole 1 mg/kg/dose BID or Omeprazole 1mg/kg/dose BID plus Ranitidine 3 mg/kg/dose BID
  Groups: Moderate/Severe Esophagitis

SUMMARY:
The goal of this study is to prospectively evaluate the impact of antacid therapy on esophagitis in children with repaired esophageal atresia. Recent clinical guidelines have attempted to define a systematic approach to the management of these patients with regards to minimizing and treating esophagitis (Krishnan et al 2016), however the quality of evidence supporting many of the recommendations are based on expert opinion or on limited, retrospective studies. Risk factors for esophagitis and optimal length of antacid therapy are not well defined. Through this study, we aim to identify risk factors for the presence of esophagitis in patients with repaired esophageal atresia. We hypothesize that antacid therapy improves esophagitis severity in children following esophageal repair.

DETAILED DESCRIPTION:
A. Specific Aims/Objectives The goal of this study is to prospectively evaluate the impact of antacid therapy on esophagitis in children with repaired esophageal atresia. Recent clinical guidelines have attempted to define a systematic approach to the management of these patients with regards to minimizing and treating esophagitis (Krishnan et al 2016), however the quality of evidence supporting many of the recommendations are based on expert opinion or on limited, retrospective studies. Risk factors for esophagitis and optimal length of antacid therapy are not well defined. Through this study, we aim to identify risk factors for the presence of esophagitis in patients with repaired esophageal atresia. We hypothesize that antacid therapy improves esophagitis severity in children following esophageal repair.

B. Background and Significance

Esophageal atresia is one of the most common congenital gastrointestinal anomalies and affects 1 in 2500 to 1 in 4000 live births (Pinheiro et al 2012; Krishnan et al 2016). Recent ESPGHAN-NASPGHAN guidelines have attempted to define a systematic approach to the post-operative management of these patients with regards to minimizing and treating esophagitis, anastomotic strictures, and feeding difficulties (Krishnan et al 2016), however the quality of evidence supporting many of the recommendations are based on expert opinion or on limited, retrospective studies. For example, there are no controlled studies describing benefit of systematic acid suppression on outcomes such as esophagitis or associated long-term sequelae such as esophageal stricture. While esophagitis in these patients has been presumed to be related to high rates of acid reflux, it is unclear that antacid therapy leads to reduced rates of esophagitis or its complications. A recent meta-analysis of four observational studies suggests that antacid therapy with PPI is not associated with lower rates of esophageal strictures (Miyake et al 2018). Boston Children's Hospital Esophageal and Airway Treatment Center has one of the largest cohorts of children with esophageal atresia in the United States with the opportunity to study the impact of antacid therapy in management of esophagitis in repaired esophageal atresia.

C. Design and Methods

Prospective analysis of inpatient and ambulatory pediatric patients and their medical records at Boston Children's Hospital who have undergone primary anastomosis repair of esophageal atresia beginning upon IRB approval.

For the remainder of the protocol, "year-1" refers to the initial set of testing/procedures/clinic visits occurring during the study period. "Year-2" refers to the second set of routine testing/procedures/clinic visits occurring approximately one year after the "year-1" time point.

Inclusion Criteria: All repaired esophageal atresia patients with primary esophageal anastomosis are eligible to enroll at the time of their routine year-1 surveillance endoscopy / pH-impedance studies:

* For patients with histology showing no or mild esophagitis, no erosive esophagitis, and reflux index <3% on pH-metry, antacid therapy will be discontinued.
* For patients with histology showing moderate or severe esophagitis and/or erosive esophagitis and/or reflux index > 3% on pH-metry, antacid therapy with PPI will be initiated. For patients already taking PPI at therapeutic dosing, an H2 blocker will be added.

Data collection will include:

* Clinical history including age at enrollment, gender, esophageal atresia type, date of esophageal atresia repair, associated anomalies, history of prematurity, history of anastomotic leak, history of prior esophageal dilations, history of gastrostomy tube placement, history of fundoplication, hiatal hernia
* Medication history
* Symptom questionnaire at enrollment and at 1 year post-enrollment
* pH-Impedance data (including reflux index, retrograde bolus movements, mean acid clearance time, mean bolus clearance time, and proximal events) at enrollment and at 1 year post-enrollment
* Endoscopic findings as well as data from interventions (e.g. dilations, injections) at enrollment and at 1 year post-enrollment
* Histology from esophageal biopsies
* Outcome data including primary outcome histologic esophagitis severity and secondary outcomes including presence of Barrett's esophagus, erosive esophagitis on endoscopy, and rates of BRUEs, respiratory infections, hospitalizations, and need for dilations

ELIGIBILITY:
Inclusion Criteria:

* All repaired esophageal atresia patients with primary esophageal anastomosis treated at Boston Children's Hospital are eligible to enroll before or at year-1 surveillance endoscopy

Exclusion Criteria:

* Patients with jejunal or colonic interpositions

Ages: 30 Days to 17 Years | Sex: All
Age Groups: Child
Study Population: Pediatric esophageal atresia patients with primary esophageal anastomosis at Boston Children's Hospital
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Esophagitis | 2 years
  Histologic esophagitis score graded as none, mild, moderate or severe

SECONDARY OUTCOMES:
Esophagitis (macroscopic) | 2 years
  Erosive esophagitis score graded according to LA classification
Barrett's esophagus | 2 years
  Presence of intestinal metaplasia (Barrett's esophagus) on esophageal biopsies
Hospitalizations | 2 years
  Need for intercurrent hospitalization for any reason

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Boston Childrens Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krishnan U, Mousa H, Dall'Oglio L, Homaira N, Rosen R, Faure C, Gottrand F. ESPGHAN-NASPGHAN Guidelines for the Evaluation and Treatment of Gastrointestinal and Nutritional Complications in Children With Esophageal Atresia-Tracheoesophageal Fistula. J Pediatr Gastroenterol Nutr. 2016 Nov;63(5):550-570. doi: 10.1097/MPG.0000000000001401. PMID 27579697
- [Background] Miyake H, Chen Y, Hock A, Seo S, Koike Y, Pierro A. Are prophylactic anti-reflux medications effective after esophageal atresia repair? Systematic review and meta-analysis. Pediatr Surg Int. 2018 May;34(5):491-497. doi: 10.1007/s00383-018-4242-4. Epub 2018 Mar 13. PMID 29536176
- [Background] Pinheiro PF, Simoes e Silva AC, Pereira RM. Current knowledge on esophageal atresia. World J Gastroenterol. 2012 Jul 28;18(28):3662-72. doi: 10.3748/wjg.v18.i28.3662. PMID 22851858